CLINICAL TRIAL: NCT05104021
Title: The Effect of Mobilization of Environmental Play on Fear and Pain Levels in the Postoperative Period Between 6-12 Years Old Children With Acute Appendicitis
Brief Title: Environmental Game After Appendicitis Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Collaborators: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Melike Yilmaz Akdag, Principal Investigator, RN, MSc, Okan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018.06.01
Record Dates: First submitted 2021-08-19; First posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Healthy
Keywords: Pain; Fear; Pediatric surgery; Game; Appendicitis
MeSH Terms: conditions — Pain; Appendicitis | interventions — Games, Experimental

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- game group (Experimental): Children who accepted to participate in the game were taken to the playground with minimum two and maximum four people. After the children were introduced to each other, the rules of the game were explained. Between the children playing, dice were rolled to determine the starting order of the game. The player who scored the highest number had the right to start the game first. With the help of the stopwatch, the playing time was started, and the children played the game in accordance with the rules.
  For the child who first reached the square of the world, the time was stopped and recorded in the "Child Follow-up Form". The game was played with a maximum game duration of 15 minutes. In the same way, the times of the children who reached the world square in the second, third and fourth places were recorded on the "Follow-up Form".
  Interventions: Device: game
- control group (No Intervention): Children in the control group were allowed to walk for 15 minutes on a flat surface in the clinic accompanied by the researcher and their parents. As soon as the child came out of his room, the time was started with the help of a stopwatch. The time was stopped when the child went back to bed.
  The pain and fear scores of each child who completed the game and mobilization were evaluated separately and simultaneously by the child, parent and researcher with the help of the "Visual Analog Scale" and the "Child Fear Scale", and then the physiological parameter measurements were made by the researcher and the "Child Follow-up Form" was evaluated after the procedure. and data collection was terminated.

INTERVENTIONS:
Device: game — The game is played with a maximum of four people. Beginning points are marked with blue, red, yellow and green colors, the game progress direction is The starting color for the player is determined with the help of arrows. Dice with the biggest number The child who throws starts the game first from the starting point that belongs to him. Play ground Each child who completes a circuit around him reads from his second point. it tries to go inwards (to the world square) in the direction it points. Equivalent to card check box The next child draws one of the face down cards. the instruction written on the back of the card.
  implements. Then he puts the card on the back of the other cards. Cards are reward (go forward), penalty (backward) git) cards. Coming second to the same frame during the game The child first starts the game from the starting point of the child in the square. First The child who manages to enter the world square wins the game.
  Arms: game group

SUMMARY:
This study was conducted to determine the effect of environmental play and mobilization on fear and pain levels of children aged 6-12 years who had acute appendicitis surgery.

DETAILED DESCRIPTION:
It was conducted with children aged 6-12 years in the postoperative period in a randomized controlled manner. Children in the intervention (n:50) group were mobilized by playing environmental games.The children in the control group (n:50) underwent routine mobilization of the clinic.

The data were collected with the "Child Follow-up Form", which was created to evaluate the child's demographic characteristics, physiological parameters, pain and fear.

ELIGIBILITY:
Inclusion Criteria:

* Being between 6-12 years old,
* Being open to communication and cooperation,
* No visual or hearing impairment,
* Appendectomy surgery,
* First mobilization after surgery.
* Parent's willingness to participate in the study can be sorted.

Exclusion Criteria:

* Having a mental or neurological disability,
* Children with hearing and vision impairment

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
The effect of environmental play on premobilization pain score of children | 30 seconds
  Visual Analog Scale (VAS) was used for determine pain level in this research. Scale got 0 to 10 points (0 (Good) to 10 (Bad)).
The effect of environmental play on the postmobilization pain score of children | 30 seconds
  Visual Analog Scale (VAS) was used for determine pain level in this research. Scale got 0 to 10 points (0 (Good) to 10 (Bad)).
The effect of environmental play on children's fear score before mobilization | 30 seconds
  Child Fear Scale (CFS) was used for determine fear score in this research. Scale got 0 to 4 points (0 (good) to 4 (bad)).
The effect of environmental play on children's fear score after mobilization | 30 seconds
  Child Fear Scale (CFS) was used for determine fear score in this research. Scale got 0 to 4 points (0 (good) to 4 (bad)).
The effect of environmental play on the pulse rate of children before mobilization | 60 seconds
  pulse rate
The effect of environmental play on the pulse rate of children after mobilization | 60 seconds
  pulse rate
The effect of environmental play on the blood pressure of children before mobilization | 60 seconds
  blood pressure
The effect of environmental play on the blood pressure of children after mobilization | 60 seconds
  blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul okan university, Tuzla, Istanbul, Turkey (Türkiye)